## <u>Preadmission Skin Wipe Use for Surgical Site Infection Prophylaxis in Adult Orthopaedic Surgery</u> <u>Patients</u>

NCT03401749 Last updated 2/23/18

A prospective observational cohort study

**Contributing Authors:** 

Eva Lehtonen<sup>1</sup> Orthopaedic Research Fellow

Sam Huntley<sup>1</sup> Medical Student

Andrew Moon<sup>1</sup> Medical Student

Sameer Naranje<sup>1</sup>
Joint Surgeon, Department of Orthopaedics

Gerald McGwin, PhD<sup>1,2</sup>, Statistician

Ashish Shah, MD<sup>1</sup>, (ashishshah@uabmc.edu) Foot and Ankle Surgeon, Primary Investigator

<sup>1</sup>Department of Orthopaedic Surgery, University of Alabama at Birmingham; Birmingham, AL

<sup>2</sup>Department of Epidemiology, University of Alabama at Birmingham; Birmingham, AL

Corresponding Author:

Ashish Shah, M.D.
Associate Professor, Director of Clinical Research
Department of Orthopaedic Surgery
1313 13th Street South, Suite 226
Birmingham, AL 35205

#### CONSENT FORM

TITLE OF RESEARCH: Efficacy of Preadmission Theraworx Wipe Use for Skin Decolonization and Surgical Site Infection Prophylaxis in Adult Orthopedic Surgery Patients: A Randomized Controlled Trial

IRB PROTOCOL NO.: IRB-300000508

**PRINCIPAL INVESTIGATOR:** Ashish Shah, M.D.

### Purpose of the Research

We are asking you to take part in a research study. This research study will test how the addition of Theraworx<sup>TM</sup> wipes or Chlorhexidine Gluconate (CHG) wipes to our standard pre- operative skin preparation effect the colonization rate of many bacteria. These bacteria are among the most common causes of surgical site infections after orthopedic surgeries. This study will also test how the addition of Theraworx<sup>TM</sup> wipes or Chlorhexidine Gluconate (CHG) wipes effects the rate of surgical site infections. We will instruct you how to use the wipes and provide you the wipes to use at home the evening before surgery. We will also provide and administer the wipes on the site of the surgery before the procedure begins. There is literature supporting that the use of Theraworx<sup>TM</sup> or CHG wipes lowers the rate of skin colonization. This is a randomized prospective study and will enroll 500 participants; all of them will come from UAB orthopaedic clinics.

#### **Explanation of Procedures**

If you enter the study, you will be placed in one of three groups:

- 1. One group will receive a standard skin preparation before your surgery. This group is the control group and will undergo orthopedic surgery following UAB's standard guidelines.
- 2. Another group will be given 2% Chlorhexidine Gluconate (CHG) wipes to take home during your last visit before the surgery. You will be given thorough instructions on how to administer the wipes the night before the surgery. Then, a nurse will use the wipe on you one hour before your standard pre-operative skin preparation on the day of the surgery.
- 3. The last group will be given Theraworx<sup>TM</sup> wipes to take home during your last visit before the surgery. You will be given thorough instructions on how to administer the wipes the night before the surgery. Then, a nurse will use the wipe on you one hour before your standard pre-operative skin preparation on the day of the surgery.

#### **Risks and Discomforts**

There may be a small chance of breach of confidentiality as a result of electronic information being hacked or stolen. You will be assigned to a group by chance, which may prove to be less effective or to have more side effects than the other study group or alternatives. Some patients may experience mild skin irritation or redness on the application site. Up to 10% may experience dryness, itching, or rash on the application site. Very rarely (less than 1% of patients), patients may experience a serious allergic reaction within minutes after the application of the wipe. Please inform your treatment team if you have ever experienced an allergic reaction to CHG or any other skin product. Symptoms of severe allergic reaction include wheezing or difficulty breathing; swelling of the face; hives that can quickly progress to more serious symptoms; severe body rash; or shock, which is a life-threatening condition that occurs when the body is not getting enough blood flow. If you experience these symptoms seek medical attention immediately.

#### **Benefits**

If you are in the group not receiving the topical wipe, you may not directly benefit from taking part in this study. However, this study may help us better understand how to decrease the positive colonization rate in the general population undergoing similar surgeries and maybe decrease post-surgical complications caused by bacterium. This study may also help raise the awareness for future investigations and possibly provide an updated option on standard skin preparation for orthopaedic surgeries.

#### **Alternatives**

Your alternative is not to participate in the study.

#### Confidentiality

Information obtained about you for this study will be kept confidential to the extent allowed by law. However, research information that identifies you may be shared with the UAB Institutional Review Board (IRB) and others who are responsible for ensuring compliance with laws and regulations related to research, including people on behalf of Dr. Ashish Shah and the Office for Human Research Protections (OHRP). The information from the research may be published for scientific purposes; however, your identity will not be given out. This consent document will be placed in your file at UAB Hospital facility. The document will become part of your medical record chart.

Your consent form will be placed in your medical record at UAB Health System or Children's of Alabama. This may include either a paper medical record or electronic medical record (EMR). An EMR is an electronic version of a paper medical record of your care within this health

system. Your EMR may indicate that you are on a clinical trial and provide the name and contact information for the principal investigator.

If you are receiving care or have received care within this health system (outpatient or inpatient) and are participating in a research study, results of research tests or procedures (i.e. laboratory tests, imaging studies and clinical procedures) may be placed in your existing medical record.

If you have never received care within this health system (outpatient or inpatient) and are participating in a research study, a medical record will be created for you to maintain results of research tests or procedures.

Results of research tests or procedures may be placed in your medical record. All information within your medical record can be viewed by individuals authorized to access the record.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### **Voluntary Participation and Withdrawal**

Whether or not you take part in this study is your choice. There will be no penalty if you decide not to be in the study. If you decide not to be in the study, you will not lose any benefits you are otherwise owed. You are free to withdraw from this research study at any time. Your choice to leave the study will not affect your relationship with this institution.

You may be removed from the study without your consent if the sponsor ends the study, if the study doctor decides it is not in the best interest of your health, or if you are not following the study rules.

If you are a UAB student or employee, taking part in this research is not a part of your UAB class work or duties. You can refuse to enroll, or withdraw after enrolling at any time before the study is over, with no effect on your class standing, grades, or job at UAB. You will not be offered or receive any special consideration if you take part in this research.

#### **Cost of Participation**

There will be no cost to you for taking part in this study. The costs of your standard medical care will be billed to you and/or your insurance company in the usual manner.

#### **Payment for Participation in Research**

You will not be paid for taking part in this study.

| Payment for Research-Related Injuries |
|---|
| UAB has not provided for any payment if you are harmed as a result of taking part in this study If such harm occurs, treatment will be provided. However, this treatment will not be provided free of charge. |

If you have any questions, concerns, or complaints about the research or a research-related injury including available treatments, you may contact Dr. Ashish Shah. He will be glad to answer any of your questions. Dr. Shah's number is 205-930-6722.

Questions

If you have questions about your rights as a research participant, or concerns or complaints about the research, you may contact the UAB Office of the IRB (OIRB) at (205) 934-3789 or toll free at 1-855-860-3789. Regular hours for the OIRB are 8:00 a.m. to 5:00 p.m. CT, Monday through Friday. You may also call this number in the event the research staff cannot be reached or you wish to talk to someone else.

| Legal Rights You are not waiving any of your legal rights by signing this informed consent document. | | | |
|---|---|---|---|
| | | Signatures | |
| | | Your signature below indicates that you have read (or been read) the info<br>above and agree to participate in this study. You will receive a copy of thi | • |
| Signature of Participant | Date | | |
| Signature of Principal Investigator or Person Obtaining Consent | Date | | |

# University of Alabama at Birmingham AUTHORIZATION FOR USE/DISCLOSURE OF PROTECTED HEALTH INFORMATION (PHI) FOR RESEARCH

| Participant Name: UAB Research Protocol: Efficacy of Preadmission Theraworx <sup>™</sup> Wipe Use | IRB Protocol Number: IRB<br>Principal Investigator: | |
|---|---|---|
| for Skin Decolonization and SSI Prophylaxis in Adult Orthopedic Surgery Patients: A Randomized Controlled Trial | | y, Division of Orthopaedics |
| What is the purpose of this form? You are being asked to sign this form so that UAB may use and release your protected health information for research. Participation in research is voluntary. If you choose to participate in the research, you must sign this form so that your protected health information may be used for the research. | | |
| Why do the researchers want my protected health information health information as part of the research protocol listed above an | | |
| What protected health information do the researchers want to limited to information and/or records of any diagnosis or treatm sexually transmitted diseases (e.g., HIV, etc.) or communicable diseidentifiers, including but not limited to your name, social security dates of service, etc.; any past, present, and future history, example reports and treatments of whatever kind, including but psychiatric/psychological treatment; financial/billing information medical bills, and any other information related to or collected whether the information was collected for research or non-research | nent of disease or condition<br>eases, drug/alcohol depend<br>y number, medical record re<br>inations, laboratory results<br>ut not limited to drug<br>n, including but not limited<br>for use in the research p | en, which may include<br>ency, etc.; all personal<br>number, date of birth,<br>s, imaging studies and<br>g/alcohol treatment,<br>ed to copies of your<br>rotocol, regardless of |
| Who will disclose, use and/or receive my protected health in informed consent documents, including but not limited to, the phaservices related to the research (whether at UAB or elsewhere); of Children's of Alabama, Eye Foundation Hospital, and the Jeffersor their operations; the IRB and its staff; the sponsor of the research and any outside regulatory agencies, such as the Food and Drug A other legal and/or regulatory functions for which access to participations. | nysicians, nurses and staff and staff and their operating units of UAI or County Department of Heal of the and its employees and agent Administration, providing on | and others performing<br>B, HSF, UAB Highlands,<br>ealth, as necessary for<br>ats, including any CRO;<br>versight or performing |
| How will my protected health information be protected once information that is given to the study sponsor will remain private sponsor is not required to follow the federal privacy laws. Ho organizations that are not required to follow federal privacy laws remain protected. | te to the extent possible, e<br>wever, once your informa | ven though the study<br>tion is given to other |
| <b>How long will this Authorization last?</b> Your authorization for Authorization does not have an expiration date. | or the uses and disclosu | res described in this |
| <b>Can I cancel this Authorization?</b> You may cancel this Author Investigator, in writing, referencing the research protocol and IRB It the study doctor and staff will not use any new health information to use the protected health information that was provide | Protocol Number. If you can<br>nation for research. Howe | cel this Authorization,<br>ever, researchers may |
| <b>Can I see my protected health information?</b> You have a right to r<br>However, to ensure the scientific integrity of the research, you w<br>until after the research protocol has been completed. | | |
| Signature of participant: | | Date: |
| or participant's legally authorized representative: | | Date: |
| Printed Name of participant's representative: | | |

Page 5 of 5 Version Date: 02/16/18

Relationship to the participant: